CLINICAL TRIAL: NCT01239446
Title: Hybrid Single-Photon Emission Computed Tomography/Computed Tomography Coronary Angiography for the Assessment of the Presence and Hemodynamic Significance of CAD in Asymptomatic Patients After Mediastinal Irradiation for Hodgkin Lymphoma.
Brief Title: Hybrid SPECT/CTCA for the Assessment of the Presence and Hemodynamic Significance of CAD in Asymptomatic Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Yafim Brodov, MD, Rambam HEalthcare Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0390-10-RMB_BRODOV
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Hodgkin Lymphoma Treated With Mediastinal Irradiation
Keywords: Hodgkin lymphoma; mediastinal irradiation; Coronary Artery Disease
MeSH Terms: conditions — Hodgkin Disease; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Not relevant (there is no intervention in the present study) — Not relevant (there is no intervention in the present study)

SUMMARY:
Mediastinal irradiation for treatment of malignancy increases the risk for coronary artery disease (CAD), while diabetes mellitus or other known risk factors can be absent at the time of the first coronary event. Radiation-induced atherosclerosis affects the coronary ostia and proximal coronary segments, or causes diffuse microvascular damage. Younger patients and those exposed to high radiation doses (> 35 Gy) have a higher risk for developing premature CAD and likely may benefit from coronary assessment.

A novel hybrid imaging technique that combines SPECT and CTCA has been shown to overcome the individual pitfalls and the diagnostic challenges of stand-alone SPECT and CCTA, improve the lesion detectability and sensitivity in patients with balanced diffuse lesions as well as the specificity and mainly PPV of CTCA.

The aim of the study is to perform hybrid SPECT/CTCA in asymptomatic patients with HL who have received radiotherapy to the mediastinum in order to allow an early diagnosis of hemodynamically significant CAD that will need further therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic HL patients without evidence of disease and without prior history of CAD that underwent mediastinal irradiation due to HL

Exclusion Criteria:

* Known CAD (these patients will be excluded from the imaging study, but will be analyzed as separate control group)
* active HL or other active malignancy
* chronic renal failure
* pregnant/ nursing women
* previous allergic reaction to iodine contrast media

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Extent of coronary artery plaques and number of perfusion defects in patients enrolled. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Healthcare Campus, Haifa, Israel